CLINICAL TRIAL: NCT00005769
Title: Hormone Replacement Therapy and Insulin Action: A Double-Blind, Parallel, Placebo-Controlled Hormone Intervention Study in Postmenopausal Women
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCRR-M01RR00109-0744; M01RR000109 (NIH)
Record Dates: First submitted 2000-06-01; First posted 2000-06-02 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: Menopause
MeSH Terms: interventions — Hormone Replacement Therapy

INTERVENTIONS:
Drug: Hormone Replacement Therapy

SUMMARY:
Considerable controversy exists regarding the effect of estrogen and progesterone on insulin sensitivity in postmenopausal women. Thus, the goal is to examine the effect of estradiol and progestin on in vivo insulin sensitivity and pathways of intracellular glucose metabolism in postmenopausal women. This will be accomplished by examining the effects of unopposed estrogen (CEE) or combination estrogen and progestin (CEE/MPA) versus placebo therapy in 30 early menopausal women (defined from 6 months to 3 years post-cessation of menses). Women will be treated for 16 weeks and the outcome measures will be: 1) insulin sensitivity and glucose oxidation as determined by euglycemic clamp, 2) assessments of insulin sensitivity on muscle biopsy cultures with the primary endpoints being glucose uptake and glycogen accumulation/synthesis, 3) protein levels of insulin action cascade steps based on muscle biopsy Western blots.

ELIGIBILITY:
Inclusion Criteria:

* 6 months to 3 years since cessation of menses
* BMD 24-33
* no surgically induced menopause

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States